CLINICAL TRIAL: NCT01930981
Title: Prospective Assessment of Associations Between Pre-transplant Comorbidities and Post-transplant Toxicities and Quality of Life
Brief Title: Associations Between Pre-transplant Comorbidities and Post-transplant Toxicities and Quality of Life
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2574.00; 4R00HL088021-03 (NIH)
Record Dates: First submitted 2013-08-15; First posted 2013-08-29 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Hematologic Malignancies; Other Diagnoses, Comorbidities, and Complications
Keywords: quality of life; toxicities; hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are interested in studying whether and how medical problems other than primary cancer before hematopoietic cell transplantation would impact the profiles of quality of life and toxicities post-transplantation for patients with blood cancers. We want to see if by assessing comorbidities (such as diabetes) early on, we can identify those patients who will have more toxicities or limitations in their quality of life after transplant. The generated information could set the stage for future intervention studies aiming to improve quality of life for patients with blood cancers after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HCT candidates who are >18 years of age
* Able to speak and read English
* Able to provide informed consent
* Access to a telephone for study-related communications
* Diagnosed with a hematological malignant disease
* Willing to complete survey packets at 5 time-points, spanning two years

Exclusion Criteria:

* HCT candidates who are 18 years or younger at the time of study enrollment
* HCT candidates who cannot read, write, or speak English
* Patients with diagnoses of non-malignant diseases, or solid tumors are primary disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hematological malignancies who are being treated with allogeneic hematopoietic cell transplantation (HCT) at the Seattle Cancer Care Alliance.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The MD Anderson Symptom Inventory | Change from Baseline in Symptoms at 3,6,12,and 24 months
  A 19-item instrument, it assesses physical symptoms and their interference with life.
The Functional Assessment of Cancer Therapy Bone Marrow Transplant Scale | Change from Baseline in Symptoms at 3,6,12,and 24 months
  A 49-item questionnaire measuring quality of life in bone marrow transplant patients, it measures physical, functional, social/family and emotional well-being in addition to bone marrow transplant-specific concerns.
The EQ-5D | Change from Baseline in Symptoms at 3,6,12,and 24 months
  This measure is used to measure utilities that can be used to calculate a quality adjusted survival score.
The Social Activity Log | Change from Baseline in Symptoms at 3,6,12,and 24 months
  This measure captures the frequency and diversity of social activities outside of daily responsibilities.
ENRICHD Social Support Instrument | Change from Baseline in Symptoms at 3,6,12,and 24 months
  This measures social support, including participation in social activities and perception of social support.
The Cancer and Treatment Distress Scale | Change from Baseline in Symptoms at 3,6,12,and 24 months
  This is a 25-item scale assessing distress related to perceived demands from events specific to cancer survivors.
The Patient Health Questionnaire-9 | Change from Baseline in Symptoms at 3,6,12,and 24 months
  The PHQ-9 measures measures depression and parallels the nine diagnostic symptom criteria of the DSM-IV for Major Depressive Disorder.

SECONDARY OUTCOMES:
National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) | at 90 days
  We will measure toxicities using the NCI CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed L Sorror, MD; MSc, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States